CLINICAL TRIAL: NCT03575429
Title: Autism Adaptive Community-based Treatment to Improve Outcomes Using Navigators (ACTION) Network
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Boston Medical Center (Other); University of Miami (Other); University of Massachusetts, Boston (Other); Kaiser Permanente (Other); Children's Hospital of Philadelphia (Other); Boston University (Other)
Responsible Party: Principal Investigator, Amy M. Wetherby, Distinguished Research Professor, Florida State University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Health Services Research
Other Study IDs: R01HD093055 (NIH)
Record Dates: First submitted 2018-06-15; First posted 2018-07-02 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Pediatrics; Social Communication; Family Navigators
MeSH Terms: conditions — Autism Spectrum Disorder; Communication

STUDY DESIGN:
Intervention Model Description: This study uses a 2-stage sequential multiple assignment randomized trial (SMART) design to optimize a menu of interventions by comparing the order and dose that best meet the needs of families. In stage 1, families will be randomly assigned to one of two study arms for 3 months. Stage 2 interventions will be for another 3 months and will be adapted based on the primary tailoring variable. Early responders will continue the same intervention and slow responders will be re-randomized to an adapted intervention for the next 3 months. The adaptations in stage 2 for slow responders include continuing the treatment arm, adding the other treatment arm, or increasing the dose of the treatment arm. Due to extenuating circumstances associated with COVID-19 from 2020-22, unplanned changes were necessary for slower recruitment than anticipated. Recruitment for the 2-stage SMART ended to allow completion of intervention and outcome measures. Recruitment continued for just stage 1 intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and diagnosticians for all measures will be kept blind to group assignment to treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Engagement Intervention (Active Comparator): Family navigators will engage families to access resources and support when they first learn their child has signs of autism spectrum disorder (ASD) using an intervention that integrates motivational interviewing (MI) and problem-solving education (PSE). The family navigator will meet with parents for up to 6 individual MI+PSE sessions for each 3-month stage of intervention.
  Interventions: Behavioral: Engagement Intervention
- Engagement + Coaching Intervention (Active Comparator): Family navigators will engage families to access resources and support when they first learn their child has signs of autism spectrum disorder (ASD) using an intervention that integrates MI+PSE. Family navigators will also coach families to embed intervention strategies for toddlers with ASD in everyday activities using the Early Social Interaction (ESI) model. ESI teaches parents how to support their child's social communication, language, play and behaviors in everyday routines, activities, and places. The family navigator will meet with parents for 12 weekly home visits for each 3-month stage of intervention.
  Interventions: Behavioral: Engagement + Coaching Intervention

INTERVENTIONS:
Behavioral: Engagement Intervention — Family navigators will use MI to engage families to decrease resistance and build motivation and commitment to challenging behavior changes by eliciting and reflecting broader goals and values, linking those values to specific behavior change, and negotiating a "menu" of options for change based on individual preferences. PSE will be used by the Family Navigators to guide families in selecting an objective, measurable problem, then proceed through a series of steps that involve goal setting, brainstorming and evaluating solutions, choosing a solution, and action planning.
  Arms: Engagement Intervention
Behavioral: Engagement + Coaching Intervention — ESI program planning entails identifying goals and objectives for the child and teaching strategies and supports for parents. Each session includes the following components: 1) setting the stage to develop that visit's agenda and gather updates; 2) intervention implementation that must include the following steps to coach the parent: a) review the objective, b) use modeling, guided/caregiver practice, or video review to teach the strategy, c) provide specific feedback to the parent, and d) problem solving and plan for next time; steps a-d are repeated for 3-5 activities per session; and 3) summarize plans for parent implementation between sessions. Families are invited to Autism Navigator How-To Guide for Families, a self-guided web-based course, with an online weekly group meeting.
  Arms: Engagement + Coaching Intervention

SUMMARY:
The Autism Adaptive Community-based Treatment to Improve Outcomes Using Navigators (ACTION) Network-a new interdisciplinary network of 6 institutions-will blend clinical effectiveness and implementation research designs to study individual and combined effects of 2 evidence-based interventions in real world settings. The first is to engage families to access resources and support when they first learn their child has signs of ASD using an evidence-based intervention that integrates motivational interviewing and problem-solving education (MI+PSE). The second is to coach families to embed evidence-based intervention strategies for toddlers with ASD in everyday activities using the Early Social Interaction (ESI) model. In Phase 1, investigators will compare the effectiveness of adaptive interventions that use MI+PSE with and without ESI on parent and child outcomes in 3 sites in Florida and Massachusetts using a 2-stage Sequential Multiple Assignment Randomized Trial (SMART) design. In Phase 2, investigators will construct an adaptive intervention to optimize the effects and study the feasibility of implementation in new sites in California. This research network can build the capacity of community-based systems to provide earlier and widespread access to cost-efficient, community-viable treatment and be ready for immediate and rapid implementation across the US.

DETAILED DESCRIPTION:
Research shows that a stable diagnosis of autism spectrum disorder (ASD) can be made by trained professionals at 18-24 months and yet the median age of diagnosis in the US is 4-5 years of age. Lower income, minority, and rural families receive a diagnosis up to 1.5 years later and more likely miss the window of opportunity for early intervention (EI). One of the greatest challenges researchers face, in spite of scientific advances and investments, is how to bridge the healthcare science-to-service gap and address health disparities in access to evidence-based EI for children with ASD. Doing this would be the best solution to improve lifelong outcomes, reduce costs to society, and change the landscape of autism.

The Autism Adaptive Community-based Treatment to Improve Outcomes Using Navigators (ACTION) Network-a new interdisciplinary network of 6 institutions-will blend clinical effectiveness and implementation research designs to study individual and combined effects of 2 evidence-based interventions in real world settings: 1) engage families to access resources and support when they first learn their child has signs of ASD using an evidence-based intervention that integrates motivational interviewing and problem solving education (MI+PSE); and 2) coach families to embed evidence-based intervention strategies for toddlers with ASD in everyday activities using the Early Social Interaction (ESI) model. Building on existing infrastructure, the Network will infuse mobile technology using the Autism Navigator® collection of web-based courses and tools.

Families will be recruited by screening in community-based primary care and EI systems in 3 diverse regions in 2 states: Florida and Massachusetts. In Phase 1, investigators will compare the effectiveness of adaptive interventions that use MI+PSE with and without ESI in a 2-stage Sequential Multiple Assignment Randomized Trial (SMART) design on family engagement in EI, parent use of intervention strategies in everyday activities, and child outcomes of social communication, active engagement, autism symptoms, developmental level, and adaptive behavior. In Phase 2, investigators will construct an adaptive intervention to optimize the effects of MI+PSE with ESI based on the SMART and study the feasibility of implementation in two new service systems in California: Kaiser Permanente Healthcare System and the National Black Church Initiative.

The ACTION Network brings a unique interdisciplinary team with expertise spanning early detection, maternal mental health, clinical trials, health disparities, implementation science, and policy. Using dynamic technology platform the Network has ambitious dissemination aims of informing a community of change agents committed to impact at the population level. This research network can build the capacity of community-based systems to provide earlier and widespread access to cost-efficient, community-viable treatment and be ready for immediate and rapid implementation across the US. Findings will advance science by providing researchers with a method for rapidly deploying evidence-based practices, enabling research at younger ages-accelerating genetic, neuroscience, and intervention research-and lead to transformative changes in workforce development and healthcare delivery.

ELIGIBILITY:
Inclusion Criteria:

* Positive screen for autism by community provider in a primary care setting
* Child is between 12 and 24 months old
* Parent completes the Smart Early Screening for Autism and Communication Disorders (ESAC)
* Parent participates in the home observation to complete the Systematic Observation of Red Flags (SORF) of ASD
* Positive autism screen on the SORF
* Lives in the designated study region in Florida and Massachusetts

Exclusion Criteria:

* Parent/caregiver declines to participate in the study
* Child is already receiving early intervention services
* Child does not screen positive for autism on the ESAC and/or SORF
* Child is over 24 months old

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Parent contingent responsiveness change over time | Baseline, 3, 6, 9, and 12 months after the start of intervention
  Parent contingent responsiveness will be periodically assessed using the Measure of Active Engagement and Transactional Supports (MAETS). The MAETS is a rating of a video-recorded home observation of parent-child interaction during everyday activities. The MAETS includes 8 components: participation and a productive role; predictable activities; language that follows the child's focus of attention; child initiations; balance of communicative turns; messages to support child comprehension; verbal and nonverbal models; and appropriate expectations and demands. Each component is scored on a 4-point scale where 0 = Absent, 1 = Emerging, 2 = Practicing, and 3 = Mastery. Total scores range from 0 to 32 and higher scores indicate that the level of parent support is better.
  Families assigned to the Engagement Intervention will be compared with families assigned to Engagement + Coaching Intervention at each time point.
Observation of DSM-5 features of autism spectrum disorder change over time | Baseline, 3, 6, 9, and 12 months after the start of intervention
  Features of autism spectrum disorder (ASD) will be periodically measured using the Systematic Observation of Red Flags (SORF) of ASD. The SORF is measured from a home observation of everyday activities. The SORF includes 11 red flags in social communication and social interaction and 11 red flags in restricted and repetitive behaviors using the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) diagnostic features rated on a 3 point scale. The total number of red flags ranges from 0 to 22 and higher scores indicate more red flags of ASD. The total composite score ranges from 0 to 66 and higher scores indicate more diagnostic features of ASD.
Child social communication change over time | Baseline, 3, 6, 9, and 12 months after the start of intervention
  Change in social communication skills will be periodically measured with the Communication and Symbolic Behavior Scales (CSBS) Behavior Sample. Interactions between the child and caregiver will be videotaped and later rated for social communication skills and converted into scores. The raw scores will be summed to form a social, speech, and symbolic composite. The social composite includes emotion and eye gaze and communication and gestures; and possible composite scores range from 0 to 64. The speech composite includes sounds and words, and possible composite scores range from 0 to 54. The symbolic composite includes understanding and object use, and possible scores for this composite range from 0 to 53. The total summed score for all 3 composites ranges from 0 to 171. Higher scores on the composites and total indicate better social communication skills.
  Families assigned to the Engagement Intervention will be compared with families assigned to Engagement + Coaching Intervention.

SECONDARY OUTCOMES:
Autism Diagnostic Observation Schedule (ADOS) | 12 months after the start of intervention
  Autism symptoms will be measured with the Autism Diagnostic Observation Schedule (ADOS), Second Edition, the gold standard diagnostic measure of ASD. The revised algorithms forming Social-Affect and Restricted Repetitive Behavior ratings of autism symptoms will be used. Scores range from 1 to 10 and higher scores indicate more autism symptoms. A total of score of 1 to 3 indicates no signs of ASD, a score of 4 or 5 suggests that the child may have ASD, while a score of 6 to 10 is indicative of ASD.
  Families assigned to the Engagement Intervention will be compared with families assigned to Engagement + Coaching Intervention.
Mullen Scales of Early Learning (MSEL) | 12 months after the start of intervention
  This study will use four scales of the Mullen Scales of Early Learning (MSEL) to measure developmental level: Fine Motor; Visual Reception; Expressive Language; and Receptive Language. The average of the four cognitive scales forms an Early Learning Composite. The 4 cognitive scales are measured with T scores that range from 10 to 90 based on a mean T score of 50. A higher T score indicates a better developmental level for the child's age. The Early Learning Composite is measured with Standard scores that range from 40 to 160 based on a mean standard score of 100. A higher standard score indicates a better developmental level for the child's age.
  Families assigned to the Engagement Intervention will be compared with families assigned to Engagement + Coaching Intervention.
Vineland Adaptive Behavior Scales (VABS-3) | 12 months after the start of intervention
  Adaptive Behavior will be measured with the Vineland Adaptive Behavior Scales, 3rd edition (VABS-3). The VABS-3 provides a standard score in four domains: Communication, Daily Living Skills, Socialization, and Motor Skills. The domain scores are averaged to form an Adaptive Behavior Composite score. The domain and composite standard scores range from 40 to 160 based on a mean standard score of 100. A higher domain and composite standard score indicates a better adaptive behavior for the child's age.
  Families assigned to the Engagement Intervention will be compared with families assigned to Engagement + Coaching Intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Wetherby, PhD, Principal Investigator — Florida State University Autism Institute
Locations (3):
- United States (3):
  - University of Miami, Coral Gables, Florida
  - Florida State University Autism Institute, Tallahassee, Florida
  - Boston Medical Center Corporation, Boston, Massachusetts